CLINICAL TRIAL: NCT00472199
Title: A Phase IV Randomised, Double-blind, Placebo-controlled, Dose Titration Trial With Pramipexole (Sifrol, Mirapexin) 0.125-0.75 mg/Day Per os to Investigate the Long-term Efficacy, Safety and Tolerability in Patients With Idiopathic Moderate to Severe Restless Legs Syndrome for 26 Weeks Followed by a 26 Week Open-label Extension Treatment Period
Brief Title: Long-term Efficacy, Safety and Tolerability of Pramipexole in Patients With Idiopathic Moderate to Severe Restless Legs Syndrome (RLS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.629; EUDRACT2006-006431-42
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2012-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pramipexole (Experimental): 4 weeks of flexible dose-titration (to optimise efficacy and tolerability), starting at 0.125 mg once daily with the potential to increase or decrease the dose in steps to 0.25 mg, 0.5 mg and 0.75 mg, with the final dose level subsequently fixed for 22 weeks.
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): 4 weeks of flexible dose-titration as for the investigational product; with the dose subsequently fixed for 22 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole
  Arms: Pramipexole
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of the current study will be the evaluation of long-term efficacy of a 26-weeks treatment with pramipexole in patients with idiopathic moderate to severe Restless Legs Syndrome (RLS) in comparison to placebo.

The key secondary objectives are to assess the effects on clinical global impressions - global improvement (CGI-I) (based on CGI-I responder rate) and on RLS (based on IRLS responder rate) for 26 weeks under pramipexole in comparison to placebo. Further secondary objectives are to investigate the incidence and severity of augmentation and rebound and to assess the effects on patient global impression (PGI) (based on PGI responder rate), on RLS symptoms (based on the RLS-6 scales), on associated mood disturbance (based on item 10 of the IRLS), on pain in limbs (based on a visual analogue scale (VAS)), on quality of life in RLS (based on Johns Hopkins RLS-QoL), on general quality of life Short Form 36 (SF-36) and on safety (based on adverse events (AE) profile) of pramipexole in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent consistent with International Conference on Harmonization - Good Clinical Practice (ICH-GCP) and local Institutional Review Board/Independent Ethics Committee (IRB/IEC) requirements obtained prior to any study procedures being performed and the ability and willingness to comply with study treatment regimen and to attend study assessments
2. Male or female out-patients aged 18-85 years
3. Diagnosis of idiopathic RLS according to the clinical RLS criteria of the International Restless Legs Syndrome Study Group (IRLSSG) [P03-03355]. All four criteria must be present to fulfil the diagnosis of RLS.
4. RLS symptoms present at least 2 to 3 days per week during the last 3 months prior to baseline (Visit 2)
5. IRLS total score >15 at baseline (Visit 2)

Exclusion Criteria:

1. Women of child-bearing potential (i.e. premenopausal women, or postmenopausal women less than 6 months after last menses) who do not use during the clinical trial an adequate method of contraception such as: double barrier protection (e.g. diaphragm or condom and spermicide), intrauterine device, hormonal therapy (oral, injectable, or subcutaneous), or partner's surgical sterilization
2. Any woman of child-bearing potential not having a negative pregnancy test at screening
3. Breastfeeding women
4. Patients with known hypersensitivity to pramipexole or any other component of the investigational product or placebo tablets
5. Diagnosis of augmentation under previous pharmacological RLS treatment
6. Concomitant or previous pharmacologic therapy as follows: Any intake of dopamine agonists within 14 days prior to baseline (Visit 2); Any intake of levodopa within 14 days prior to baseline (Visit 2); Unsuccessful prior treatment with non-ergot dopamine agonists (e.g. pramipexole, ropinirole);

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (42):
- Austria (2):
  - 248.629.4302 Boehringer Ingelheim Investigational Site, Innsbruck
  - 248.629.4304 Boehringer Ingelheim Investigational Site, Linz
- 248.629.3201 Boehringer Ingelheim Investigational Site, Edegem, Belgium
- Finland (5):
  - 248.629.35801 Boehringer Ingelheim Investigational Site, Espoo
  - 248.629.35805 Boehringer Ingelheim Investigational Site, Helsinki
  - 248.629.35804 Boehringer Ingelheim Investigational Site, Joensuu
  - 248.629.35802 Boehringer Ingelheim Investigational Site, Oulu
  - 248.629.35806 Boehringer Ingelheim Investigational Site, Tampere
- Germany (9):
  - 248.629.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 248.629.4908 Boehringer Ingelheim Investigational Site, Bochum
  - 248.629.4901 Boehringer Ingelheim Investigational Site, Ellwangen
  - 248.629.4904 Boehringer Ingelheim Investigational Site, Hellersdorf
  - 248.629.4906 Boehringer Ingelheim Investigational Site, Herborn
  - 248.629.4905 Boehringer Ingelheim Investigational Site, Leipzig
  - 248.629.4909 Boehringer Ingelheim Investigational Site, Schwerin
  - 248.629.4903 Boehringer Ingelheim Investigational Site, Steglitz
  - 248.629.4907 Boehringer Ingelheim Investigational Site, Würzburg
- Ireland (3):
  - 248.629.35301 Boehringer Ingelheim Investigational Site, Carrigtohill
  - 248.629.35302 Boehringer Ingelheim Investigational Site, Co. Kildare
  - 248.629.35303 Boehringer Ingelheim Investigational Site, Co. Tipperary
- Netherlands (6):
  - 248.629.31001 Boehringer Ingelheim Investigational Site, Bennebroek
  - 248.629.31005 Boehringer Ingelheim Investigational Site, Hoogwoud
  - 248.629.31006 Boehringer Ingelheim Investigational Site, Musselkanaal
  - 248.629.31002 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 248.629.31003 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 248.629.31004 Boehringer Ingelheim Investigational Site, Rijswijk
- Slovakia (5):
  - 248.629.4204 Boehringer Ingelheim Investigational Site, Bratislava
  - 248.629.4205 Boehringer Ingelheim Investigational Site, Bratislava
  - 248.629.4202 Boehringer Ingelheim Investigational Site, Brezno
  - 248.629.4201 Boehringer Ingelheim Investigational Site, Košice
  - 248.629.4203 Boehringer Ingelheim Investigational Site, Martin
- Spain (5):
  - 248.629.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 248.629.3405 Boehringer Ingelheim Investigational Site, Granada
  - 248.629.3401 Boehringer Ingelheim Investigational Site, Madrid
  - 248.629.3403 Boehringer Ingelheim Investigational Site, San Sebastián
  - 248.629.3406 Hospital Arnau de Vilanova, Valencia
- United Kingdom (6):
  - 248.629.44003 Boehringer Ingelheim Investigational Site, Chorley
  - 248.629.44006 Boehringer Ingelheim Investigational Site, Edgbaston, Birmingham
  - 248.629.44004 Boehringer Ingelheim Investigational Site, Glasgow
  - 248.629.44001 Boehringer Ingelheim Investigational Site, Manchester
  - 248.629.44002 Boehringer Ingelheim Investigational Site, Reading
  - 248.629.44005 Boehringer Ingelheim Investigational Site, Waterloo, Liverpool

REFERENCES:
- See also: Related Info — http://trials.boehringer-ingelheim.com/content/dam/internet/opu/clinicaltrial/com_EN/results/248/248.629_Literature.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 331 patients enrolled, 329 were treated with study drug. Two patients were randomized, but before their first intake of trial medication they decided to not participate in the study.
Groups:
- Pramipexole: 4 weeks of flexible dose-titration (to optimise efficacy and tolerability), starting at 0.125 mg once daily with the potential to increase the dose to 0.25mg and to further increase or decrease the dose in steps to 0.5 mg and 0.75 mg, with the final dose level subsequently fixed for 22 weeks. mode of administration: Oral, once daily in the evening (2 to 3 hours before bedtime) form: tablets
- Placebo: 4 weeks of flexible dose-titration as for the investigational product; with the dose subsequently fixed for 22 weeks. mode of administration: Oral, once daily in the evening (2 to 3 hours before bedtime) form: tablets
Period: Overall Study
Arm/Group | Pramipexole | Placebo
Started | 166 | 163
Completed | 131 | 103
Not Completed | 35 | 60
Not completed — Adverse Event | 19 | 23
Not completed — Lack of Efficacy | 4 | 25
Not completed — Lost to Follow-up | 2 | 4
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 6 | 5
Not completed — personal reason | 0 | 1
Not completed — patient was asymptomatic | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole | Placebo | Total
Number analyzed (Participants) | 166 | 163 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12.7) | 55.8 (11.4) | 56.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 94 | 196
  Male | 64 | 69 | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLS) Total Score After 26 Weeks
Description: IRLS total score ranging from 0 (no RLS symptoms) to 40 (very severe RLS symptoms)
Time Frame: Baseline and 26 weeks
Population: Intent to treat analysis. Number of randomized patients with a baseline and at least one non-missing post-baseline measure. Imputation by last observation carried forward (LOCF) for post-baseline values
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
Scores on a scale | -13.7 (0.8) | -11.1 (0.8)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Analysis of covariance for changes from baseline with factors treatment and country and using baseline as covariate; Test type: Superiority or Other; p = 0.0077, ANCOVA; Mean Difference (Net) = -2.6, 95% CI [-4.6 to -0.7], Standard Error of Mean 1

2. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Responder Rate
Description: CGI-I scores ranging from '1' (very much improved) to '7' (very much worse), CGI-I responder have scoring 1 or 2 (at least much improved)
Time Frame: after 26 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
participants
  CGI-I responder (at least much improved) | 111 | 80
  CGI-I non-responder | 51 | 79
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel

3. Secondary Outcome: International Restless Legs Syndrome (IRLS) Study Group Rating Scale Responder Rate
Description: IRLS response was defined as at least 50% reduction in IRLS total score from baseline. IRLS total score ranging from 0 (no RLS symptoms) to 40 (very severe symptoms)
Time Frame: after 26 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
participants
  IRLS responder | 95 | 68
  IRLS non-responder | 67 | 91
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0044, Cochran-Mantel-Haenszel

4. Secondary Outcome: Patient Global Impression (PGI) Responder Rate
Description: PGI scores ranging from '1' (very much better) to '7' (very much worse), PGI responder have scoring 1 or 2 (at least much better)
Time Frame: after 26 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
participants
  PGI responder (much better or very much better) | 101 | 70
  PGI non-responder | 61 | 89
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0011, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in Restless Legs Syndrome-6 (RLS-6) Score "Satisfaction With Sleep" After 26 Weeks
Description: The score is an 11-point Likert scale, ranging from "none/not at all" (0) to "very severe" (10), to reflect the patient's condition during the previous week
Time Frame: baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
Scores on a scale | -2.5 [-5.0 to 0.0] | -2 [-4.0 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0489, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.0, 95% CI [-1.1 to -0.9]

6. Secondary Outcome: Change From Baseline in RLS-6 Score "Severity Falling Asleep" After 26 Weeks
Description: as for outcome 5
Time Frame: Baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
Scores on a scale | -3 [-5.0 to 0.0] | -1 [-4 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0315, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.0 to 0.0]

7. Secondary Outcome: Change From Baseline in RLS-6 Score "Severity During the Night" After 26 Weeks
Description: The question was rated on an 11-point Likert scale, ranging from "none/not at all" (0) to "very severe" (10), to reflect the patient's condition during the previous week
Time Frame: baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
Scores on a scale | -3 [-5.0 to 0.0] | -2 [-5.0 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0735, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.0 to 0.0]

8. Secondary Outcome: Change From Baseline in RLS-6 Score "Severity During the Day When at Rest" After 26 Weeks
Description: as for outcome 5
Time Frame: Baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
Scores on a scale | -3 [-5.0 to 0.0] | -1 [-4.0 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.8410, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.0 to 0.0]

9. Secondary Outcome: Change From Baseline RLS-6 Score "Severity During the Day Engaged in Activities" After 26 Weeks
Description: as for outcome 5
Time Frame: Baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
Scores on a scale | 0 [-1.0 to 0.0] | 0 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.9241, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.0 to 0.0]

10. Secondary Outcome: Change From Baseline in RLS-6 Score "Tired or Sleepy During the Day" After 26 Weeks
Description: as for outcome 5
Time Frame: Baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
Scores on a scale | -1 [-3.0 to 0.0] | -1 [-3.0 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.8093, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.0 to 0.0]

11. Secondary Outcome: Change From Baseline in IRLS Mood Disturbance Score (Item 10) After 26 Weeks
Description: Mood disturbance associated with RLS symptoms ranging from 0 (none) to 4 (very severe)
Time Frame: Baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 159
scores on a scale | -1 [-2.0 to 0.0] | -1 [-2.0 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0583, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.0 to 0.0]

12. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score for Pain in Limbs After 26 Weeks
Description: The scale measures pain on a continuous 100 mm axis ranging from no pain (0 mm) to unbearable pain (100 mm)
Time Frame: Baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 162 | 158
Scores on a scale | -26 [-47.0 to -5.0] | -15 [-46.0 to 0.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0916, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -5.0, 95% CI 2-sided [-5.5 to -4.5]

13. Secondary Outcome: Change From Baseline in Quality of Life in RLS (RLS QoL) Score After 26 Weeks
Description: RLS QoL total score ranging from 0 to 100 with higher values indicating better quality of life
Time Frame: Baseline and 26 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 157 | 153
Scores on a scale | 15 [5.0 to 25.0] | 12.5 [2.5 to 27.5]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.5905, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.5, 95% CI 2-sided [2.2 to 2.8]

14. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Dimension Bodily Pain After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating less bodily pain
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 157 | 152
Scores on a scale | 12 [0.0 to 31.0] | 9 [-1.0 to 24.5]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0179, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.0, 95% CI 2-sided [1.6 to 2.4]

15. Secondary Outcome: Change From Baseline in SF-36 Dimension General Health After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating better health status
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 155 | 152
Scores on a scale | 0 [-5.0 to 10.0] | 0 [-5.0 to 10.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.5450, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2.0, 95% CI 2-sided [1.7 to 2.3]

16. Secondary Outcome: Change From Baseline in SF-36 Dimension Mental Health After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating better mental health
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 155 | 152
Scores on a scale | 5 [-5.0 to 15.0] | 5 [-5.0 to 10.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.1456, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.3 to 0.3]

17. Secondary Outcome: Change From Baseline in SF-36 Dimension Physical Functioning After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating better physical functioning
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 156 | 152
Scores on a scale | 0 [0.0 to 10.0] | 0 [-5.0 to 10.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.2915, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]

18. Secondary Outcome: Change From Baseline in SF-36 Dimension Role Limitations Due to Emotional Problems After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating less limitations due to emotional problems
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 156 | 152
Scores on a scale | 0 [-8.3 to 16.7] | 0 [0.0 to 16.7]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.3131, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]

19. Secondary Outcome: Change From Baseline in SF-36 Dimension Role Limitations Due to Physical Problems After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating less limitations due to physical problems
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 156 | 152
Scores on a scale | 6.3 [0.0 to 18.8] | 6.3 [0.0 to 18.8]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.5713, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]

20. Secondary Outcome: Change From Baseline in SF-36 Dimension Social Functioning After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating better social functioning
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 157 | 152
Scores on a scale | 0 [0.0 to 12.5] | 0 [0.0 to 25.0]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.8432, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]

21. Secondary Outcome: Change From Baseline in SF-36 Dimension Vitality After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating better vitality
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 155 | 152
Scores on a scale | 6.3 [0.0 to 18.8] | 3.1 [-6.3 to 12.5]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0206, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 6.3, 95% CI 2-sided [5.9 to 6.6]

22. Secondary Outcome: Change From Baseline in SF-36 Dimension Mental Component Summary After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating better health
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 155 | 152
Scores on a scale | 1.7 [-2.4 to 8.3] | 1.9 [-2.3 to 6.7]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.5602, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.6, 95% CI 2-sided [0.4 to 0.8]

23. Secondary Outcome: Change From Baseline in SF-36 Dimension Physical Component Summary After 26 Weeks
Description: Score ranging from 0 to 100 with higher scores indicating better health
Time Frame: Baseline and 26 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 155 | 152
Scores on a scale | 2.1 [-0.5 to 7.5] | 2 [-2.0 to 5.9]
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.1360, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.0, 95% CI 2-sided [0.8 to 1.1]

24. Secondary Outcome: Diagnosis of Classified Augmentation According to Independent Expert Panel
Description: Augmentation is a worsening of RLS symptoms and may manifest as increased severity and the involvement of other extremities or as a shift of RLS symptoms to a time period that is 2 or more hours earlier than was typical of the time of symptom onset during the initial course of beneficial stable treatment or the state before recently starting treatment.
Time Frame: after at least 4 weeks of treatment
Population: Treated Set and where patients received study medication for at least 4 weeks (Treated Set includes all patients who were documented to have taken at least one dose of of treatment)
Measure: Number; unit: participants
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 152 | 149
participants | 18 | 14

25. Secondary Outcome: Worsening of RLS Symptoms (by at Least 4 Points in the IRLS Total Score Compared to Baseline) After Treatment Discontinuation
Description: Worsening of RLS symptoms, in comparison to baseline, following abrupt treatment discontinuation (for patients with no added RLS therapy after study drug discontinuation).
  Assessment of worsening of RLS was based on the IRLS total score assessed 7 ± 1 days after treatment discontinuation (the end of the study or premature discontinuation) compared with that at baseline. Analysis considered the number of patients experiencing a clinically relevant deterioration of ≥4 points in total IRLS score 7 ± 1 days after discontinuation of trial medication compared with baseline.
Time Frame: after at least 1 week of treatment discontinuation
Population: Treated Set, all patients who were documented to have taken at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 135 | 133
participants | 14 | 2
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Superiority or Other; p = 0.0022, Mantel Haenszel

26. Secondary Outcome: Baseline, Week 26 Mean Supine Systolic Blood Pressure
Time Frame: Baseline, Week 26
Population: Treated Set, all patients who were documented to have taken at least one dose of study medication
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 166 | 163
mm Hg
  Baseline | 133.4 (16.9) | 132.7 (18.4)
  Week 26 | 132.3 (16.4) | 132.2 (16.5)

27. Secondary Outcome: Baseline, Week 26 Mean Standing Systolic Blood Pressure
Time Frame: Baseline, Week 26
Population: Treated Set, all patients who were documented to have taken at least one dose of study medication
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 166 | 163
mm Hg
  Baseline | 132.6 (17.3) | 130.6 (18.2)
  Week 26 | 132.4 (18.2) | 130.1 (17.1)

28. Secondary Outcome: Baseline, Week 26 Mean Supine Diastolic Blood Pressure
Time Frame: Baseline, Week 26
Population: Treated Set, all patients who were documented to have taken at least one dose of study medication
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 166 | 163
mm Hg
  Baseline | 79.2 (9.7) | 79.6 (9.7)
  Week 26 | 78.3 (9.7) | 79.5 (9.4)

29. Secondary Outcome: Baseline, Week 26 Mean Standing Diastolic Blood Pressure
Time Frame: Baseline, Week 26
Population: Treated Set, all patients who were documented to have taken at least one dose of study medication
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 166 | 163
mm Hg
  Baseline | 82.7 (10.5) | 81.7 (10.7)
  Week 26 | 80.5 (10.6) | 80.8 (10.0)

30. Secondary Outcome: Baseline, Week 26 Mean Supine Pulse Rate
Time Frame: Baseline, Week 26
Population: Treated Set, all patients who were documented to have taken at least one dose of study medication
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 166 | 163
bpm
  Baseline | 68.5 (9.6) | 68.7 (10.6)
  Week 26 | 69.1 (8.9) | 68.3 (10.6)

31. Secondary Outcome: Baseline, Week 26 Mean Standing Pulse Rate
Time Frame: Baseline, Week 26
Population: Treated Set, all patients who were documented to have taken at least one dose of study medication
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 166 | 163
bpm
  Baseline | 74.6 (10.2) | 74.0 (10.7)
  Week 26 | 74.1 (8.9) | 75.0 (10.6)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Pramipexole | Placebo
Serious Adverse Events (participants affected / at risk) | 8/166 | 3/163
Other Adverse Events (participants affected / at risk) | 70/166 | 58/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=166) | Placebo (N=163)
Appendicitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=166) | Placebo (N=163)
Nausea (Gastrointestinal disorders) | 24 | 6
Fatigue (General disorders) | 18 | 15
Headache (Nervous system disorders) | 13 | 17
Restless legs syndrome (Nervous system disorders) | 11 | 11
Somnolence (Nervous system disorders) | 11 | 8
Nasopharyngitis (Infections and infestations) | 7 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.